CLINICAL TRIAL: NCT00268671
Title: Phase I/II Trial of Weekly Docetaxel and Cisplatin for Locoregional Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Docetaxel in Squamous Cell Carcinoma of the Head and Neck (TAX + Cisplatin in SCCHN)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976G_2501
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
Study Objectives:

* To determine the MTD (maximal tolerated dose) and recommended dose of a weekly docetaxel and cisplatin combination regimen for locoregional recurrent/metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
* To determine the response rate of the recommended dose
* To determine the safety and tolerability of the recommended dose

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (of original primary tumor) locoregional recurrent and/or metastatic following prior radiotherapy and/or surgery and not amenable to further curative local therapy for SCCHN
* Measurable disease as defined by at least the longest diameter measured as 20 mm by conventional CT or 10 mm by spiral CT. Physical measurements are allowed if longest diameter is 20 mm by caliper measurements.
* ECOG performance status 0-2
* Adequate bone marrow and hepatic function as evidenced by the following:

  * Hematology (Bone marrow):

    * Neutrophils ≥ 1.50 x 10^9/L
    * Platelets ≥ 100 x 10^9/L
    * Hemoglobin ≥ 10 g/dL
  * Hepatic function:

    * AST and/or ALT: < 2X ULN (Upper Limit of Normal)
    * Bilirubin < 1X ULN
* Adequate renal function with calculated or measured glomerular filtration rate of > 60 ml/min calculated by the Cockcroft- Gault method
* No severe intercurrent illness or other serious illness or medical conditions including but not limited to:

  * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry.
  * Active uncontrolled infection
  * Active peptic ulcer
  * Chronic obstructive pulmonary disease requiring hospitalization during the year preceding study entry
* No prior chemotherapy for recurrent/advanced SCCHN with platinum or taxane regimen (primary radiosensitizing platinum allowed).
* No other diagnosed malignancy other than basal cell carcinoma of the skin or cervix carcinoma in situ

Exclusion Criteria:

* Prior therapy with taxanes either adjuvant, neoadjuvant, concurrent or in advanced stage disease
* Prior chemotherapy for locoregional recurrent/metastatic SCCHN with palliative intent
* Contraindications from

  * the medical history (i.e. known hepatitis, HIV) and physical exam
  * laboratory tests (hematology, biochemistry)
  * 12-lead electrocardiogram
  * blood pressure and pulse
* Pregnancy
* Breast-feeding
* Treatment with any investigational product in the last 4 weeks before study entry
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Presence or sequelae of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* History of hypersensitivity to the study drug(s) or to drugs with a similar chemical structure
* Impaired hepatic function, as shown by bilirubin greater than upper limits of normal and/or AST greater than 2 times upper limits of normal
* Impaired renal function, as shown by measured or calculated creatinine clearance of < 60 ml/min or absolute creatinine level > 1.5 upper limit of normal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04

PRIMARY OUTCOMES:
AE SAE collection | from the inform consent signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Monique Furlan, Study Director — Sanofi